CLINICAL TRIAL: NCT05216835
Title: A Phase I/II Open-label, Multi-center Study to Assess Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of AZD7789, an Anti-PD-1 and Anti-TIM-3 Bispecific Antibody, in Patients With Relapsed or Refractory Classical Hodgkin Lymphoma.
Brief Title: Safety and Preliminary Efficacy Assessment of AZD7789 in Patients With Relapsed or Refractory Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9571C00001; 2021-003569-36 (EudraCT Number)
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Relapsed or Refractory Classical Hodgkin Lymphoma
Keywords: Pharmacokinetics; Classical Hodgkin Lymphoma (cHL); Dose Expansion; Dose escalation; r/r cHL; programmed cell death protein-1 (PD-1); Accelerated titration design (ATD); T cell immunoglobulin and mucin domain-containing protein-3 (TIM-3); Modified toxicity probability interval-2 (mTPI-2); Bispecific antibody; Immunotherapy
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Dose Escalation (Experimental): Patients with anti-PD-1/PD-L1 exposed r/r cHL will receive sabestomig to determine the recommended phase 2 dose (RP2D).
  Interventions: Drug: Sabestomig (AZD7789)
- Cohort B1: Dose Expansion (Experimental): Patients with anti-PD-1/PD-L1 exposed r/r cHL will receive sabestomig once the RP2D has been determined.
  Interventions: Drug: Sabestomig (AZD7789)
- Cohort B2: Dose Expansion (Experimental): Patients with anti-PD-1/PD-L1 naïve r/r cHL will receive sabestomig once the RP2D has been determined.
  Interventions: Drug: Sabestomig (AZD7789)

INTERVENTIONS:
Drug: Sabestomig (AZD7789) — Patients will receive sabestomig (PD-1/TIM-3 bispecific monoclonal antibody) via intravenous infusion.

SUMMARY:
The study is intended to assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of sabestomig (AZD7789) in patients with relapsed/refractory classical Hodgkin Lymphoma (r/r cHL).

DETAILED DESCRIPTION:
This is a Phase I/II, open-label multi-center study will have sabestomig administered via intravenous infusion on Cycle 1 Day 1 to adult/young adult patients with relapsed/refractory classical Hodgkin Lymphoma (r/r cHL). This study will have 2 parts: Phase 1 (Part A) Dose Escalation and Phase 2 (Part B) Dose Expansion.

Patients will be treated with study intervention for a maximum of 35 cycles, or until disease progression, unacceptable toxicity, withdrawal of consent, or if other reasons to discontinue treatment occur.

The trial was intended to be Phase I/II trial (but the trial never moved forward to Phase 2). Hence, the study Phase was updated to Phase I.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 16 years of age at the time of obtaining informed consent
* Eastern Cooperative Oncology Group performance status of 0 or 1 at screening
* At least one positron emission tomography (PET)-avid measurable lesion according to Modified Lugano Criteria after the last line of therapy.
* Confirmed histological diagnosis of active relapse/refractory cHL
* Failed at least 2 prior lines of systemic therapy.
* No previous treatment with anti-TIM-3.
* Adequate organ and bone marrow function
* Non-pregnant women and willingness of female patients to avoid pregnancy or male participants willing to avoid fathering children through highly effective methods of contraception
* Minimum body weight ≥ 40 kg for all participants.

Exclusion Criteria:

* Unresolved toxicities of ≥ Grade 2 from prior therapy
* Any prior ≥ Grade 3 imAE while receiving prior checkpoint inhibitor immunotherapy
* Patients with central nervous system (CNS) involvement or leptomeningeal disease.
* History of allogeneic stem cell transplant or organ transplantation.
* Any venous or arterial thromboembolic event within ≤ 6 months prior to the first dose of study intervention.
* Active infection including Tuberculosis (TB), human immunodeficiency virus (HIV), hepatitis A, chronic or active hepatitis B, chronic or active hepatitis C, active COVID-19 infection
* History of arrhythmia which is requires treatment, symptomatic or uncontrol led atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia
* Uncontrolled intercurrent illness.
* Active or prior documented pathologically confirmed autoimmune or inflammatory disorders.
* Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD
* Other invasive malignancy within 2 years prior to screening
* Congenital long QT syndrome or history of QT prolongation associated with other medications that cannot be changed or discontinued based on a cardiologist assessment
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose of study intervention
* Any concurrent chemotherapy, radiotherapy, investigational, biologic, or hormonal therapy for cancer treatment.

Ages: 16 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - Research Site, Duarte, California
  - Research Site, Miami, Florida
  - Research Site, Rochester, Minnesota
  - Research Site, New York, New York
  - Research Site, Houston, Texas
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Research Site, København Ø, Denmark
- Research Site, Lille, France
- Italy (2):
  - Research Site, Bologna
  - Research Site, Napoli
- Research Site, Valencia, Spain
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9571C00001&attachmentIdentifier=facc246c-51a1-409b-9b50-7764ab4a0942&fileName=CSR_Synopsis_19_Dec_2024_D9571C00001_Final_Redacted_19Feb2025_watermark.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9571C00001&attachmentIdentifier=ca82868a-2ad5-4cad-bd7d-8d4760d75c48&fileName=d9571c00001-sap-ed-3_Final_Redacted_19Feb2025_watermark.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9571C00001&attachmentIdentifier=82ae7214-584d-4a02-9082-4f4ae1210c07&fileName=_Protocol_Main_5_07May2024_English__D9571C00001_Public_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study from 18 March 2022 (First subject in) and the analyses presented in this results form are based on a final data cut-off (DCO) of 30 August 2024.
Pre-assignment Details: Participants who met the inclusion criteria and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment.
  Part B was not initiated, therefore, no participant was enrolled and analyzed for this part of the study.
Groups:
- Cohort A1: Participants with relapsed or refractory classical Hodgkin Lymphoma (r/r cHL) previously treated with anti-programmed cell death protein-1/programmed cell death-ligand 1 (anti-PD-1/PD-L1) based therapy received 2mg of sabestomig.
- Cohort A2: Participants with r/r cHL previously treated with anti-PD-1/PD-L1 based therapy received 7mg of sabestomig.
- Cohort A3: Participants with r/r cHL previously treated with anti-PD-1/PD-L1 based therapy received 22.5mg of sabestomig.
- Cohort A4: Participants with r/r cHL previously treated with anti-PD-1/PD-L1 based therapy received 75mg of sabestomig.
- Cohort A5: Participants with r/r cHL previously treated with anti-PD-1/PD-L1 based therapy received 225mg of sabestomig.
- Cohort A6: Participants with r/r cHL previously treated with anti-PD-1/PD-L1 based therapy received 750mg of sabestomig.
- Cohort A7: Participants with r/r cHL previously treated with anti-PD-1/PD-L1 based therapy received 1500mg of sabestomig.
- Cohort A8: Participants with r/r cHL previously treated with anti-PD-1/PD-L1 based therapy received 2000mg of sabestomig.
Period: Overall Study
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Started | 1 | 1 | 1 | 1 | 5 | 12 | 12 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 1 | 5 | 12 | 12 | 12
Not completed — Ongoing as of DCO (30 Aug 2024) | 0 | 0 | 0 | 0 | 3 | 10 | 10 | 9
Not completed — Death | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Study terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received any amount of study intervention.
Groups:
- Cohort A1: Participants with r/r cHL previously treated with anti-PD-1/PD-L1 based therapy received 2mg of sabestomig.
- Total: Total of all reporting groups
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 12 | 12 | 12 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | NA (NA) — Mean was not reported due to concerns with participant's confidentiality. Standard deviation was not calculable for a single participant. | NA (NA) — Mean was not reported due to concerns with participant's confidentiality. Standard deviation was not calculable for a single participant. | NA (NA) — Mean was not reported due to concerns with participant's confidentiality. Standard deviation was not calculable for a single participant. | NA (NA) — Mean was not reported due to concerns with participant's confidentiality. Standard deviation was not calculable for a single participant. | 45.8 (17.6) | 44.4 (16.0) | 38.6 (14.5) | 52.1 (21.2) | 44.0 (17.4)
Sex/Gender, Customized [Count of Participants; unit: Participants] — For single participant in a particular gender, the data was not reported under specific category, rather a customized option was used, and the data was reported as 'All' to maintain participant's confidentiality.
  Participants
    Female | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 6 | 14
    Male | 0 | 0 | 0 | 0 | 2 | 9 | 10 | 6 | 27
    All | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — For single participant in a particular ethnicity, the data was not reported under specific category, rather a customized option was used, and the data was reported as 'Other' to maintain participant's confidentiality.
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 0 | 0 | 0 | 0 | 3 | 12 | 10 | 10 | 35
    Missing | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 5
    Other | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part A (Dose Escalation): Number of Participants With Adverse Events (AEs)
Description: The safety and tolerability of sabestomig in participants with r/r cHL were assessed.
Time Frame: From start of treatment [Cycle 1 Day 1 (C1D1) (each cycle was 28 days)] up to 90 days post last dose (approximately 2 years 5 months)
Population: Safety set included all participants who received any amount of study intervention.
  CTCAE = Common Terminology Criteria for Adverse Events (version 5.0)
  1. = As assessed by the investigator.
  2. = AE of special interest derivations were programmed based on sponsor assessment of AE terms.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 12 | 12 | 12
Participants
  Any AE | 1 | 1 | 1 | 1 | 4 | 12 | 10 | 12
  Any AE possibly related to Sabestomig [a] | 0 | 1 | 0 | 1 | 3 | 10 | 8 | 6
  Any AE of CTCAE grade 3 or higher | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 2
  Any AE of CTCAE grade 3 or higher, possibly related to Sabestomig [a] | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
  Any AE with outcome = death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Any AE with outcome = death, possibly related to Sabestomig [a] | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE (including events with outcome = death) | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 0
  Any SAE (including events with outcome = death), possibly related to Sabestomig [a] | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
  Any SAE leading to discontinuation of Sabestomig | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Any SAE leading to discontinuation of Sabestomig, possibly related to Sabestomig [a] | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of Sabestomig | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  Any AE leading to discontinuation of Sabestomig, possibly related to Sabestomig [a] | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Any AE leading to cycle delay | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 3
  Any AE leading to cycle delay, possibly related to Sabestomig [a] | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Any AE of special interest [b] | 0 | 1 | 0 | 1 | 2 | 8 | 7 | 5
  Any AE of special interest [b] also considered as an immune-mediated AE [a] | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2
  Any AE of special interest [b], possibly related to Sabestomig [a] | 0 | 1 | 0 | 1 | 2 | 6 | 4 | 2
  Any AE of special interest [b] also an immune-mediated AE, possibly related to Sabestomig [a] | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2
  Any immune-mediated AE [a] | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3
  Any immune-mediated AE, possibly related to Sabestomig [a] | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3

2. Other Pre Specified Outcome: Part A (Dose Escalation): Number of Participants With Adverse Events of Special Interest (AESIs)
Description: The safety and tolerability of sabestomig in participants with r/r cHL were assessed.
  An AESI was an AE of scientific and medical interest specific to understanding of a study intervention and may have required close monitoring and rapid communication to AstraZeneca by the Investigator.
  The AESIs for sabestomig include events with a potential inflammatory or immune-mediated mechanism and which may require more frequent monitoring and/or interventions such as steroids, immunosuppressants and/or hormone replacement therapy.
Time Frame: From start of treatment [C1D1 (each cycle was 28 days)] up to 90 days post last dose (approximately 2 years 5 months)
Population: Safety set included all participants who received any amount of study intervention.
  AE of special interest derivations were programmed based on sponsor assessment of AE terms.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 12 | 12 | 12
Participants | 0 | 1 | 0 | 1 | 2 | 8 | 7 | 5

3. Primary Outcome: Part A (Dose Escalation): Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLT was defined as any ≥Grade 3 AE as per NCI CTCAE version 5 unless unequivocally due to underlying malignancy or an extraneous cause.
  The following conditions were considered as DLTs:
  * Any death not clearly due to the underlying disease or extraneous causes
  * Grade 4 imAE or anemia
  * Any ≥Grade 3 non-infectious pneumonitis or colitis of any duration
  * Specific liver transaminase elevation as per protocol
  * Any Grade 3 imAE, including rash, pruritus, or diarrhea, that does not downgrade to Grade 2 or less within 7 days
  * Grade 3 nausea, vomiting, or diarrhea that does not resolve to Grade 2 or less within 3 days of getting maximal supportive care
  * ≥Grade 3 neutropenia, without fever or systemic infection, that does not improve by at least one grade within 7 days
  * Grade 4 thrombocytopenia for more than 7 days or ≥Grade 3 thrombocytopenia along with Grade ≥2 bleeding
  * Grade 4 Cytokine Release Syndrome (CRS) of any duration or Grade 3 CRS not improving to Grade ≤2 within 72 hours
Time Frame: From first dose (C1D1) until 28 days for each participant [within 28 days DLT period]
Population: Safety set included all participants who received any amount of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 11 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Part B (Dose Expansion): Cohort B1: Objective Response Rate (ORR)
Description: The anti-tumor activity of sabestomig in participants with r/r cHL was planned to be assessed.
  ORR was defined as the percentage of participants with an objective response [Best Overall Response of a complete response (CR) or partial response (PR)] as per modified Lugano criteria (Lugano 2014), with the denominator defined as the number of participants in the response-evaluable analysis set.
  Disease response was planned to be assessed according to Blinded Independent Central Review using modified Lugano criteria (Lugano 2014).
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Groups:
- Part B: Participants with anti-PD-1/PD-L1 exposed r/r cHL were planned to receive sabestomig once the RP2D had been determined.
Arm/Group | Part B
Number analyzed (Participants) | 0

5. Primary Outcome: Part B (Dose Expansion): Cohort B2: Complete Response Rate (CRR)
Description: The anti-tumor activity of sabestomig in participants with r/r cHL was planned to be assessed.
  The CRR was defined as the percentage of participants with a CR as per modified Lugano criteria (Lugano 2014), with the denominator defined as the number of participants in the response-evaluable analysis set.
  Disease response was planned to be assessed according to Blinded Independent Central Review using modified Lugano criteria (Lugano 2014).
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

6. Primary Outcome: Part B (Dose Expansion): Number of Participants With AEs
Description: The safety and tolerability of sabestomig in participants with r/r cHL was planned to be assessed.
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

7. Secondary Outcome: Part A (Dose Escalation): Complete Response Rate (CRR)
Description: The anti-tumor activity of sabestomig in participants with r/r cHL was assessed.
  The CRR was defined as the percentage of participants with a CR as per modified Lugano criteria (Lugano 2014) as assessed by the Investigator, with the denominator defined as the number of participants in the response-evaluable analysis set.
  Disease response was assessed according to Investigator assessment using modified Lugano criteria (Lugano 2014).
Time Frame: From start of treatment [C1D1 (each cycle was 28 days)] until first documented disease progression, or last evaluable assessment in the absence of progression (up to 2 years 5 months)
Population: Response-evaluable set included all dosed participants who had measurable disease at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 12 | 12 | 12
Percentage of participants | NA — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in Statistical analysis plan (SAP). | NA — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | 0 | 33.3 | 0 | 0

8. Secondary Outcome: Part A (Dose Escalation): Objective Response Rate (ORR)
Description: The anti-tumor activity of sabestomig in participants with r/r cHL was assessed.
  The ORR was defined as the percentage of participants with an objective response (Best Overall Response of CR or PR) as per modified Lugano criteria (Lugano 2014), as assessed by the Investigator, with the denominator defined as the number of participants in the response-evaluable analysis set.
  Disease response was assessed according to Investigator assessment using modified Lugano criteria (Lugano 2014).
Time Frame: From start of treatment [C1D1 (each cycle was 28 days)] until progression, or last evaluable assessment in the absence of progression (up to 2 years 5 months)
Population: Response-evaluable set included all dosed participants who had measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 12 | 12 | 12
Percentage of participants | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | 0.0 [NA to NA] — Here, 'NA' indicated that the upper and lower limit of confidence interval did not cross the 50% probability of ORR. | 50.0 [21.1 to 78.9] | 25.0 [5.5 to 57.2] | 16.7 [2.1 to 48.4]

9. Secondary Outcome: Part A (Dose Escalation): Duration of Response (DoR)
Description: The anti-tumor activity of sabestomig in participants with r/r cHL was assessed.
  The DoR was defined as the time from the date of first documented objective response (CR or PR), as assessed by Investigator, using the modified Lugano criteria (Lugano 2014), until the date of first documented disease progression or death (by any cause in the absence of disease progression).
  Disease response was assessed according to Investigator assessment using modified Lugano criteria (Lugano 2014).
Time Frame: From first documented response until date of first documented disease progression or death from any cause, or data cut-off or end of study (whichever came first, assessed up to 2 years 5 months)
Population: Response-evaluable set included all dosed participants who had measurable disease at baseline.
  Number of participants analyzed were number of participants with objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 6 | 3 | 2
Months | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. |  | NA [2.7 to NA] — Here, 'NA' indicated that the median and lower limit of confidence interval did not cross the 50% probability of DoR. | 7.7 [7.1 to NA] — Here, 'NA' indicated that the lower limit of confidence interval did not cross the 50% probability of DoR. | 6.3 [NA to NA] — Here, 'NA' indicated that the upper and lower limit of confidence interval did not cross the 50% probability of DoR.

10. Secondary Outcome: Part A (Dose Escalation): Duration of Complete Response (DoCR)
Description: The anti-tumor activity of sabestomig in participants with r/r cHL was assessed.
  The DoCR was defined as the time from first documented CR, as per modified Lugano criteria (Lugano 2014) as assessed by the Investigator, until the date of first documented relapse/progression or death due to any cause (in the absence of disease progression).
  Disease response was assessed according to Investigator assessment using modified Lugano criteria (Lugano 2014).
Time Frame: From first documented complete response until date of first documented disease progression or death from any cause, or data cut-off or end of study (whichever came first, assessed up to 2 years 5 months)
Population: Response-evaluable set included all dosed participants who had measurable disease at baseline.
  Number of participants analyzed were number of participants with complete response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Months |  |  |  |  |  | NA [NA to NA] — Here, 'NA' indicated that data (DOCR) was not calculable due to low number of responders with CR events, as pre-specified in SAP. |  |

11. Secondary Outcome: Part A (Dose Escalation): Progression-free Survival (PFS)
Description: The anti-tumor activity of sabestomig in participants with r/r cHL was assessed.
  PFS was defined as the time from first dose until the earlier of the date of first documented disease progression, as per modified Lugano criteria (Lugano 2014) as assessed by the Investigator, or death (by any cause in the absence of disease progression or subsequent anticancer treatment).
  Disease response was assessed according to Investigator assessment using modified Lugano criteria (Lugano 2014).
Time Frame: From start of treatment [C1D1 (each cycle was 28 days)] until date of first documented disease progression or data cut-off or end of study (whichever came first, assessed up to 2 years 5 months)
Population: Full analysis set included all participants who received any amount of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 12 | 12 | 12
Months | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | 1.9 [1.4 to NA] — Here, 'NA' indicated that the lower limit of confidence interval did not cross the 50% probability of PFS. | 4.8 [2.4 to 11.9] | 5.7 [1.8 to NA] — Here, 'NA' indicated that the lower limit of confidence interval did not cross the 50% probability of PFS. | 2.1 [1.6 to 8.1]

12. Secondary Outcome: Part A (Dose Escalation): Overall Survival (OS)
Description: The anti-tumor activity of sabestomig in participants with r/r cHL was assessed.
  The OS was defined as the time from the start of treatment until death due to any cause regardless of whether participant withdraws from treatment or receives another anti-lymphoma therapy.
Time Frame: From start of treatment [C1D1 (each cycle was 28 days)] until date of death due to any cause or data cut-off or end of study (whichever came first, assessed up to 2 years 5 months)
Population: Full analysis set included all participants who received any amount of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 12 | 12 | 12
Months | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [NA to NA] — Here, 'NA' indicated that data were not analyzed due to presence of single participant during analysis as pre-specified in SAP. | NA [1.4 to NA] — Here, 'NA' indicated that the median and lower limit of confidence interval did not cross the 50% probability of OS. | NA [NA to NA] — Here, 'NA' indicated that the median and confidence interval did not cross the 50% probability of OS. | NA [NA to NA] — Here, 'NA' indicated that the median and confidence interval did not cross the 50% probability of OS. | NA [8.4 to NA] — Here, 'NA' indicated that the median and lower limit of confidence interval did not cross the 50% probability of OS.

13. Secondary Outcome: Part A (Dose Escalation): Number of Participants With Positive Anti-drug Antibodies (ADA) Against Sabestomig in Serum
Description: The presence of ADA for sabestomig in treated participants with r/r cHL was assessed.
Time Frame: On C1D1, C2D1, and until end of study [up to 2 years 5 months (each cycle was 28 days)]
Population: Immunogenicity analysis set included all participants who received at least 1 dose of study intervention with at least 1 reportable immunogenicity measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 12 | 12 | 12
Participants
  ADA prevalence | 1 | 0 | 0 | 0 | 3 | 4 | 4 | 2
  Treatment-induced ADA positive | 1 | 0 | 0 | 0 | 3 | 4 | 3 | 2
  Treatment-boosted ADA | 1 | 0 | 0 | 0 | 3 | 3 | 4 | 2
  ADA incidence | 1 | 0 | 0 | 0 | 3 | 4 | 4 | 2
  ADA positive at baseline and at least one post-baseline | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ADA positive at baseline and not positive at post-baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ADA transient positive | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0
  ADA persistently positive | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 2

14. Secondary Outcome: Part A (Dose Escalation): Maximum Observed Concentration (Cmax)
Description: The Cmax of sabestomig in participants with r/r cHL was assessed.
Time Frame: From C1D1 [before start of infusion (SOI) and at end of infusion (EOI)] to end of study [up to 2 years 5 months (each cycle was 28 days)]
Population: Pharmacokinetic (PK) set included all participants who received at least 1 dose of study intervention with at least 1 reportable concentration.
Measure: Median (Full Range); unit: microgram (ug)/milliliter (mL)
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 12 | 11 | 11
microgram (ug)/milliliter (mL) | NA [0.14 to 0.14] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | NA [1.41 to 1.41] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | NA [5.80 to 5.80] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | NA [15.40 to 15.40] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | 52.49 [39.60 to 82.90] | 256.00 [172.00 to 430.00] | 516.00 [364.00 to 1480.00] | 695.10 [323.00 to 1400.00]

15. Secondary Outcome: Part A (Dose Escalation): Area Under the Concentration-time Curve (AUC)
Description: The AUC of sabestomig in participants with r/r cHL was assessed.
Time Frame: From C1D1 (before SOI and at EOI) to end of study [up to 2 years 5 months (each cycle was 28 days)]
Population: PK set included all participants who received at least 1 dose of study intervention with at least 1 reportable concentration.
Measure: Median (Full Range); unit: Day*ug/mL
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 5 | 11 | 11 | 11
Day*ug/mL |  | NA [4.24 to 4.24] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | NA [28.50 to 28.50] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | NA [88.80 to 88.80] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | 273.00 [110.00 to 518.00] | 2256.00 [1710.00 to 4780.00] | 4687.00 [2740.00 to 8370.00] | 6883.00 [2560.00 to 8120.00]

16. Secondary Outcome: Part A (Dose Escalation): Clearance (CL)
Description: The CL of sabestomig in participants with r/r cHL was assessed.
Time Frame: From C1D1 (before SOI and at EOI) to end of study [up to 2 years 5 months (each cycle was 28 days)]
Population: as for outcome 15
Measure: Median (Full Range); unit: Liter (L)/Day
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 4 | 11 | 9 | 11
Liter (L)/Day |  | NA [1.3200 to 1.3200] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | NA [0.7210 to 0.7210] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | NA [0.8160 to 0.8160] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | 0.4925 [0.2910 to 1.9800] | 0.2321 [0.1030 to 0.4200] | 0.2211 [0.1010 to 0.3180] | 0.2149 [0.1280 to 0.7020]

17. Secondary Outcome: Part A (Dose Escalation): Terminal Elimination Half-life (t½λz)
Description: The t½λz of sabestomig in participants with r/r cHL was assessed.
Time Frame: From C1D1 (before SOI and at EOI) to end of study [up to 2 years 5 months (each cycle was 28 days)]
Population: as for outcome 15
Measure: Median (Full Range); unit: Day
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 4 | 11 | 9 | 11
Day |  | NA [2.880 to 2.880] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | NA [8.980 to 8.980] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | NA [4.730 to 4.730] — Here, 'NA' indicated that median value was not calculated for a single participant as pre-specified in the SAP. | 9.136 [3.100 to 25.000] | 12.720 [6.680 to 42.800] | 16.440 [11.200 to 22.600] | 12.070 [5.990 to 21.000]

18. Secondary Outcome: Part B (Dose Expansion): Duration of Response (DoR)
Description: The DoR of sabestomig in participants with r/r cHL was planned to be assessed.
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

19. Secondary Outcome: Part B (Dose Expansion): Duration of Complete Response (DoCR)
Description: The DoCR of sabestomig in participants with r/r cHL was planned to be assessed.
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

20. Secondary Outcome: Part B (Dose Expansion): Progression-free Survival (PFS)
Description: The anti-tumor activity of sabestomig in participants with r/r cHL was planned to be assessed.
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

21. Secondary Outcome: Part B (Dose Expansion): Overall Survival (OS)
Description: The anti-tumor activity of sabestomig in participants with r/r cHL was planned to be assessed.
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

22. Secondary Outcome: Part B (Dose Expansion): Number of Participants With Positive ADA Against Sabestomig in Serum
Description: The presence of ADA for sabestomig in treated participants with r/r cHL was planned to be assessed.
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

23. Secondary Outcome: Part B (Dose Expansion): Maximum Observed Concentration (Cmax)
Description: The Cmax of sabestomig in participants with r/r cHL was planned to be assessed.
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

24. Secondary Outcome: Part B (Dose Expansion): Area Under the Concentration-time Curve (AUC)
Description: The AUC of sabestomig in participants with r/r cHL was planned to be assessed.
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

25. Secondary Outcome: Part B (Dose Expansion): Terminal Elimination Half-life (t½λz)
Description: The t½λz of sabestomig in participants with r/r cHL was planned to be assessed.
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

26. Secondary Outcome: Part B (Dose Expansion): Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: Proportion of participants reporting different levels of presence/magnitude/interference (as applicable) of diarrhea, rash, and fatigue over time based on PRO-CTCAE was planned to be evaluated.
  PRO-CTCAE was a PRO measurement system developed to evaluate symptomatic toxicity in participants on cancer clinical trials. The PRO-CTCAE Item Library included 124 items representing 78 symptomatic toxicities drawn from the CTCAE. PRO-CTCAE items were planned to evaluate the symptom attributes of frequency, severity, interference, amount, presence/absence. Each symptomatic AE was planned to be assessed by 1 to 3 attributes. Conditional branching logic was planned to be used with electronic data capture, thereby reducing respondent burden. The recall period was planned as the past 7 days and PRO-CTCAE responses were planned to score from 0 to 4 (or 0/1 for absent/present).
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

27. Secondary Outcome: Part B (Dose Expansion): Pediatric Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (Peds-PRO-CTCAE)
Description: Proportion of participants reporting different levels of presence/magnitude/interference (as applicable) of diarrhea, rash, and fatigue over time based on peds-PRO-CTCAE was planned to be evaluated.
  The pediatric module included 130 items representing 62 symptomatic toxicities and permitted self-reporting by children and adolescents aged 7 to 17 years. In this study, 17 symptomatic toxicities were planned for selection. Thus, the total number of questions that participants would have answered ranged from 17 (assuming that no branching questions were triggered, ie, the participant answered '0' to the initial question for each symptom) to 42 items (assuming that all possible branching questions were triggered for every symptom posed to the participant).
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

28. Secondary Outcome: Part B (Dose Expansion): Patient Global Impression of Treatment Tolerability (PGI-TT)
Description: Proportion of participants reporting different levels of overall side-effect bother over time based on the PGI-TT was planned to be evaluated.
  For adult participants only, the PGI-TT item was included to assess how a participant perceived the overall burden of treatment-related side effects of cancer treatment over the past 7 days. Participants were planned to be asked to choose the response that best described the level of burden by the side effect of their cancer treatment over the past week. The planned response options were:"not at all", "a little bit", "somewhat", "quite a bit", and "very much".
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

29. Secondary Outcome: Part B (Dose Expansion): European Organization for Research and Treatment of Cancer (EORTC) Item List (IL)XX QL2 [2-item Global Health-related Quality of Life (HRQoL)]
Description: Proportion of participants reporting different levels of quality of life/health over time based on the European Organization for Research and Treatment of Cancer Item List (EORTC) ILXX QL2 items was planned to be evaluated.
  EORTC QLQ-C30 was a 30-item self-administered questionnaire designed for all cancer types. Questions were grouped into 5 multi-item functional scales (physical, role, emotional, cognitive, and social), 3 multi-item symptom scales (fatigue, pain, and nausea/vomiting), 2-item global HRQoL (QL2) scale, 5 single items assessing additional symptoms commonly reported by participants with cancer (dyspnea, loss of appetite, insomnia, constipation, and diarrhea), and 1 item on the financial impact of the disease. Participants were planned to answer QLQ-C30 questions in reference to how they had been over the past week. Final scores were planned to transform to range from 0 to 100, where higher scores indicated better functioning, better HRQoL, or greater level of symptoms.
Time Frame: Up to approximately 2 years 90 days
Population: Part B was not initiated, therefore, no participant was enrolled and analyzed for this outcome measure.
Arm/Group | Part B
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From start of treatment [Cycle 1 Day 1 (C1D1) (each cycle was 28 days)] up to 90 days post last dose (approximately 2 years 5 months)
Description: Safety set included all participants who received any amount of study intervention.
Arm/Group | Cohort A1 | Cohort A2 | Cohort A3 | Cohort A4 | Cohort A5 | Cohort A6 | Cohort A7 | Cohort A8
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 1/1 | 1/5 | 1/12 | 1/12 | 1/12
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 3/5 | 3/12 | 4/12 | 2/12
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 4/5 | 12/12 | 10/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1 (N=1) | Cohort A2 (N=1) | Cohort A3 (N=1) | Cohort A4 (N=1) | Cohort A5 (N=5) | Cohort A6 (N=12) | Cohort A7 (N=12) | Cohort A8 (N=12)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exertional rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1 (N=1) | Cohort A2 (N=1) | Cohort A3 (N=1) | Cohort A4 (N=1) | Cohort A5 (N=5) | Cohort A6 (N=12) | Cohort A7 (N=12) | Cohort A8 (N=12)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute graft versus host disease in skin (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 4 (5) | 0 (0)
Intention tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Secondary cerebellar degeneration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (3) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Part A (dose escalation) of this study was completed and Part B (dose expansion) of this study was not initiated and therefore, data were not collected and analyzed for Part B of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca.

DOCUMENTS (2):
  • Study Protocol (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT05216835/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT05216835/SAP_001.pdf